CLINICAL TRIAL: NCT05292781
Title: CHOICES for Sickle Cell Reproductive Health: Randomized Clinical Trial (RCT) of a Preconception Intervention Model for a Single Gene Disorder
Brief Title: CHOICES3: Sickle Cell Disease Parenting CHOICES
Acronym: CHOICES3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB201803021; R01HG011927 (NIH); PRO00035017 (Other: UFIRST)
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease; Sickle Cell Trait
MeSH Terms: conditions — Anemia, Sickle Cell; Sickle Cell Trait

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHOICES (Experimental): Experimental arm: receives the web-based reproductive education for individuals with sickle cell disease or sickle cell trait
  Interventions: Other: CHOICES
- eBook (electronic-Book) (Sham Comparator): Control arm with eBook education focused on sickle cell disease and sickle cell trait.
  Interventions: Other: eBook

INTERVENTIONS:
Other: CHOICES — An innovative web application to provide interactive information about reproductive health options for people with SCD or SCT. CHOICES is a multimedia intervention that provides targeted and tailored information for participants to become informed ns about their reproductive health options. Targeted to their sex and tailored to their SC reproductive health knowledge, reproductive health behavior during the previous 6 mo, and parenting plan (e.g., intention to have child with SCD or not), CHOICES presents information about options to help the participant achieve their parenting plan through reproductive partner selection based on sickle cell status, prenatal testing, ovum and sperm donation, advanced reproductive technologies, and options to avoid pregnancy or adopt. The website will be housed on secure University of Florida (UF) servers and accessible via computers or mobile devices (e.g., tablets, smart phones); device capture will inform plans for long-term dissemination.
  Arms: CHOICES
Other: eBook — e-Book contains information typically shared in clinical SCD care, including stick figure representation of inheritance because the investigator considers it unethical to withhold this basic information. It does not include other information related to the SCKnowIQ knowledge items or any of the behaviors needed to implement a parenting plan. Although not as long as CHOICES, the e-Book is sufficiently long, attractive, and engaging to retain participants randomized to the usual care control group; key factors for an adequate control condition. Interestingly, during the study and in interviews after the study, many e-Book participants commented that they were pleased to be assigned to the intervention group (they had not), which indicates that the control condition is sufficient for its intent--2-yr longitudinal retention of the sample. Also, human contact is the same for both groups, and the time-on-task on the computer is unlikely to influence study knowledge and behavior endpoints.
  Arms: eBook (electronic-Book)

SUMMARY:
The study will use web-based data collection (SCKnowIQ) and intervention delivery strategies enhanced by nudges and tailored boosters in a sample of 430 adult men and women, aged 18-45 yr with SCD (Sickle Cell Disease) or SCT (Sickle Cell Trait), at-risk, and planning within 2 years to have a child free of SCD.

DETAILED DESCRIPTION:
In a 2-year, randomized, longitudinal, repeated measures, controlled trial in 430 at-risk young adults with SCD (50%) or SCT (50%) to compare the effects of e-Book (electronic-Book) and CHOICES interventions on knowledge and behaviors across time (baseline, immediate posttest, 6, 12, 18, 24 months). The study will provide boosters tailored to knowledge deficits at 6 and 12 months and add monthly reinforcement nudges toward concordant behavior during the first 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SCD (HbSS, HbSC (Hemoglobin Sickle C Disease), HbS-beta-0 thalassemia, and HbS-beta+ thalassemia) or report of SCT (SCD is Hgb electrophoresis confirmed; SCT evaluated by SickleScan);
* Able and intends to conceive a child in the next 2 years (first child or another child);
* Speaks and reads English;
* 18 to 45 years;
* At-risk for having a child with SCD (i.e., sexual/ reproductive partner has SCD, SCT, or unknown sickle cell status); and
* Wants to avoid the risk of a child with SCD.
* The age range is based on typical reproductive age for SCD where median survival is 42 years for men and 48 years for women.

Exclusion Criteria:

* Legally blind;
* Physically unable to complete the study questionnaires or the intervention;
* Report health history of hysterectomy, tubal ligation, medically or surgically induced menopause, or vasectomy that would
* Prevent ability to bear children;
* Report a desire to remain childless or have no further children;
* Report knowing or being a relative or friend of a participant previously enrolled in the study, or
* Previous participation in a CHOICES study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 506 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Sickle Cell Reproductive Health Knowledge | Baseline up to 24 months
  Knowledge. The Sickle Cell Reproductive Health Knowledge Questionnaire measures knowledge of the genetic transmission of SCD and SCT, etiology of SCD, parenting options for people with SCD or SCT, types of contraceptives safe for people with SCD or SCT, and risks of complications during pregnancy for the woman with SCD. Responses are multiple choice options. Scores are totaled across all items, ranging from 0 to 17; higher scores reflect better knowledge than lower scores.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Wilkie, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No